CLINICAL TRIAL: NCT04263961
Title: SHERLOCk: an Integrative Genomic Approach to Solve tHe Puzzle of sevERe earLy-Onset COPD
Brief Title: An Integrative Genomic Approach to Solve tHe Puzzle of sevERe earLy-Onset COPD
Acronym: SHERLOCk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Maarten van den Berge, PhD, MD, University Medical Center Groningen
Other Study IDs: 201600328
Record Dates: First submitted 2016-04-22; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease; Severe Early-Onset COPD; SEO-COPD
Keywords: Severe Early-Onset COPD (SEO-COPD); Genotyping; Phenotyping; Susceptibility
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Disease, Chronic Obstructive, Severe Early-Onset; Disease Susceptibility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — The aim of this study is to identify why a subset of COPD patients develops such a severe COPD at early age and with relatively few packyears smoking. This will need a functional genomics approach integrating both whole genome DNA sequencing data in blood and transcriptomics data in the bronchial epithelium as well as epigenetic regulation. This will identify novel common and rare genetic variants, genes, miR's, and DNA methylation sites that contribute to severe early-onset COPD.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD GOLD I - II: Inclusion for mild-moderate COPD patients (n = 100):
  * Age between 45-65 years.
  * GOLD classification I or II according to the Global initiative for Chronic Obstructive Lung Disease (GOLD) criteria (post bronchodilator FEV1/FVC <0.7) [2].
  * Cessation of smoking for ≥6 months.
  * ≥5 packyears of smoking.
  * Absence of asthma.
  * Written informed consent.
- Controls: Inclusion for healthy controls (n = 100):
  * Age between 45-65 years.
  * Absence of COPD according to the Global initiative for Chronic Obstructive Lung Disease (GOLD) criteria (post bronchodilator FEV1/FVC <0.7) [2].
  * Cessation of smoking for ≥6 months.
  * ≥5 packyears of smoking.
  * Absence of asthma.
  * Written informed consent.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is characterized by a chronic airflow limitation associated with an abnormal inflammatory response of the airways to inhaled noxious particles or gases. It is the third leading cause of death worldwide, accounting for approximately 3 million deaths each year and the prevalence is predicted to increase even further during the coming decade (WHO 2015). In the last two decades, there has been a disappointing lack of fundamental breakthroughs in the understanding of the pathophysiology of COPD and there is currently no pharmacological treatment available that halts its relentless progression. A clear alternative for describing COPD does not exist either, while the identification of subgroups of COPD patients based on clinical, genomic and epigenomic factors would be useful. A clinically relevant phenotype with high potential of having a genetic cause is severe early-onset COPD (SEO-COPD), defined by severe airflow obstruction (FEV1 ≤ 40% predicted) at a relatively young age (≤53 years) [1]. In the UMCG, we have a continuous flow of severe COPD patients who are referred to our hospital for bronchoscopic lung volume reduction treatment or lung transplantation. Approximately 40-50% of these patients fulfil the criteria for SEO-COPD. As part of a previously approved study ("Phenotyping in COPD", METc 2014/102), these patients are routinely characterized when they are willing to participate in this study and gave their written informed consent. Characterization is performed using lung function (i.e. spirometry, body box), clinical (i.e. questionnaires, physical examination, measurement of waist-hip ratio), radiologic (HRCT-scan) and systemic parameters (venous blood collection). Moreover, the following additional samples are being extracted: bronchial biopsies, bronchial brushes and nasal brushes.

There are two objectives this study adds. The primary objective is to identify the genetic and epigenetic mechanisms underlying SEO-COPD by using the bronchial brushes and biopsies that are already extracted from the SEO-COPD patients. The secondary objective is to add two control groups (i.e. mild-moderate COPD group and healthy non-COPD control group) matched for age and smoking habits (all COPD patients referred for BLVRT or lung transplantation are ex-smokers).

Hopefully, this will eventually explore COPD susceptibility and its genetic cause, resulting in a more tailored treatment of this COPD subset.

DETAILED DESCRIPTION:
2. INTRODUCTION AND RATIONALE

2.1 Chronic Obstructive Pulmonary Disease Chronic obstructive pulmonary disease (COPD) is a common preventable and treatable disease, yet without a cure. It is characterized by persistent airflow limitation that is usually progressive and associated with an enhanced chronic inflammatory response in the airways and the lungs to noxious particles or gases [2]. COPD is a leading cause of morbidity and is estimated to become the fourth leading cause of death worldwide in 2030 [3] and results in an economic and social burden that is both substantial and increasing [2]. The diagnosis of COPD is based on the presence of airflow limitation (i.e. forced expiratory volume in 1 second (FEV1) and forced vital capacity). However, the degree of airflow limitation itself does not adequately describe the complexity of COPD because significant heterogeneity exists between patients with respect to clinical presentation, physiology, imaging, response to therapy, decline in lung function and survival. Currently, a clear alternative for describing COPD does not exist but the identification of subgroups of COPD, based on clinical factors (phenotypes), eventually extended by biomarkers reflecting underlying pathophysiological processes can be attractive. This may lead to better insights in the heterogeneity of COPD and the underlying mechanisms.

2.2 The phenotype of severe early-onset COPD Several reviews have proposed that potential phenotypes can be based on clinical manifestations, physiological manifestations, radiologic characterization, COPD exacerbations, systemic inflammation and comorbidities [4-6]. Clinical manifestations include age, smoking history, sex, ethnicity, body composition, exacerbation frequency and dyspnea level. Physiologic manifestations include amongst others lung function, decrease in lung function over time (FEV1), lung volumes, hyperinflation, hyperresponsiveness exercise capacity and muscle function. Radiologic characterization includes computed tomography (CT) scanning of the lung and for example measures of airway wall thickness or emphysema scores. Clusters of patients with similar characteristics may constitute a phenotype and can be based on expert opinion, or statistical techniques like an unsupervised cluster analysis.

A phenotype of particular clinical relevance is a subset of smokers who will develop severe COPD at an early age and with relatively few packyears smoking. In 1998, Silverman et al. defined this phenotype by severe airflow obstruction (i.e. Forced Expiratory Volume in 1 second (FEV1) <40% predicted) and age ≤53 years [1]. This severe early-onset COPD accounts for a significant part of the total personal, societal and economic burden attributed to COPD. However, despite the clinical relevance of this group of COPD patients, this definition of severe early-onset COPD is only based on FEV1 and age. Therefore, this perhaps out-dated definition lacks other phenotypical parameters, i.e. smoking history, slope of lung function decline, radiologic characterization such as emphysema, and other possible factors contributing to this phenotype. This proposed study will evaluate different phenotypes of SEO-COPD, linking it with genotypical characterization.

2.3 The genotype of severe early-onset COPD Although it is widely accepted that smoking is the main risk factor for COPD, only 20-30% of smokers will ultimately develop the disease [1]. A small subset of smokers will develop severe COPD at an early age and with relatively few packyears smoking. The question arises as to why these patients are particularly susceptible to the adverse effects of smoking. In this context, the findings of Silverman et al. are of particular interest, showing that smoking first- degree relatives of these severe early-onset COPD patients had a significantly lower FEV1 than controls of the same age and smoking habits, suggesting genetic factors to play a role in COPD development [1]. The latter is in line with findings of case-control and twin studies and it is estimated that 40-60% of the risk for development of COPD is genetically determined [7,8]. Thus far, little is known about the origins and underlying mechanisms that drive the development of severe early-onset COPD. With this proposed study, we will explore these mechanism using new possibilities for genotyping.

2.4 New possibilities for genotyping GWAS studies have identified several genetic variants associated with susceptibility to develop COPD [9-11]. Although these studies have generated important new insights, their biological interpretation has been limited. Variants that were identified so far are estimated to explain only a small percentage (approximately 8%) of the total genetic risk attributed to COPD [12]. It is important to realize that the genotyping platforms used in GWAS studies so far mainly included common SNP's, i.e. those with a minor allele frequency (MAF) >5%, whereas rare variants with a MAF <5% have been heavily underrepresented. The latter is important, since rare variants are likely to be involved in SEO-COPD. One well-known example of a rare genetic variant that is functionally related to SEO-COPD is the non- synonymous SNP in the region coding for SERPINA1 causing alpha-1-antitrypsin deficiency [13,14]. Although important, alpha-1-antitrypsin deficiency is present in only a small percentage of patients leaving a large proportion of heritability of SEO-COPD unexplained. This proposed study will include rare variants, now a feasible approach with recent advances in high-throughput whole-genome sequencing technologies [15].

2.5 Severe early-onset COPD patients referred to the UMCG Many patients with severe COPD are being referred to the University Medical Center Groningen (UMCG) every year from the entire Netherlands for a consultation on lung transplantation (LTX) or bronchoscopic lung volume reduction therapy (BLVRT) (approximately 250 per year) [16,17]. BLVRT is only performed in our center in the Netherlands. As part of a previously approved study ("Phenotyping in COPD", METc 2014/102), patients with severe COPD who are referred for BLVRT or lung transplantation are characterized when they are willing to participate and gave their written informed consent. Characterization is performed using lung function (i.e. spirometry, body box), clinical (i.e. questionnaires, physical examination, measurement of waist-hip ratio), radiologic (HRCT-scan) and systemic parameters (venous blood collection). Moreover, the following additional samples are being extracted: bronchial biopsies, bronchial brushes and nasal brushes.

There are two objectives this study adds. The primary objective is to identify the genetic and epigenetic mechanisms underlying SEO-COPD by using the bronchial brushes and biopsies that are already extracted from the SEO-COPD patients. The secondary objective is to add two control groups (i.e. mild-moderate COPD group and healthy non-COPD control group) matched for age and smoking habits (all COPD patients referred for BLVRT or lung transplantation are ex-smokers), which is currently missing.

Hopefully, this will eventually elucidate COPD susceptibility and its genetic cause, resulting in a more tailored treatment of this COPD subset.

Primary Objective:

- To identify the genetic and epigenetic mechanisms underlying SEO-COPD by using bronchial brushes and biopsies and assess how these SEO-COPD patients differ from two control groups (mild-moderate COPD and non-COPD subjects).

Secondary Objectives:

To:

* determine which common and rare genetic variants are likely causally related to the development and/or excessive progression of the disease.
* assess which COPD-associated genes and gene-networks are controlled by miR's (micro-RNA's) and DNA methylation sites.

ELIGIBILITY:
Inclusion for mild-moderate COPD patients (n = 100):

* Age between 45-65 years.
* GOLD classification I or II according to the Global initiative for Chronic Obstructive Lung Disease (GOLD) criteria (post bronchodilator FEV1/FVC <0.7) [2].
* Cessation of smoking for ≥6 months.
* ≥5 packyears of smoking.
* Absence of asthma.
* Written informed consent.

Inclusion for healthy controls (n = 100):

* Age between 45-65 years.
* Absence of COPD according to the Global initiative for Chronic Obstructive Lung Disease (GOLD) criteria (post bronchodilator FEV1/FVC <0.7) [2].
* Cessation of smoking for ≥6 months.
* ≥5 packyears of smoking.
* Absence of asthma.
* Written informed consent.

4.3 Exclusion criteria

Exclusion for both mild-moderate COPD patients and healthy controls:

* Subjects must be able to adhere to the study visit schedule and other protocol requirements.
* Presence of acute infections (such as hepatitis, pneumonia, pyelonephritis) in the previous 3 months.
* Signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic or cerebral disease.
* Malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
* Known recent substance abuse.
* Females of childbearing potential without an efficient contraception.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: With the previously approved study ("Phenotyping in COPD", METc 2014/102), a large cohort of ex-smoking SEO-COPD patients (n = 150) is already being assembled, and therefore not part of the protocol.
  Important for this study; we will recruit 100 ex-smoker, mild-moderate COPD patients (COPD GOLD I-II) and 100 non-COPD controls matched for age, gender, and smoking status who smoked a similar number of packyears.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Common and rare genetic variants that contribute to severe early-onset COPD | 1 day
  Difference in gene expression between those who develop COPD and those who do not after smoking about the same amount of packyears.

SECONDARY OUTCOMES:
Spirometry | 1 day
  Spirometry
Bronchial hyperresponsiveness | 1 day
  BHR-test
Bodybox, diffusion | 1 day
  Body-box
Clinical parameters | 1 day
  Comorbidity
Clinical parameters - Questionnaires | 1 day
  St. Georges
Radiologic parameters | 1 day
  High-resolution computed tomography (HR-CT)
Systemic parameters | 1 day
  Blood levels Assessing the systemical parameters of 100 healthy controls to compare with those of the 150 SEO-COPD patients (linked with primary outcome).
Histological parameters | 1 day
  Biopsies
Immunological parameters | 1 day
  air liquid interface

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - UMCG, Groningen